CLINICAL TRIAL: NCT05088213
Title: Suction Mini-PCNL Versus Standard PCNL for the Management of 2-4cm Kidney Stones: An International Multi-centre Randomized Controlled Trial
Brief Title: Suction Mini-PCNL Versus Standard PCNL for the Management of 2-4cm Kidney Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Aceves of Wake Forest University Medical Center (Unknown); University College London Hospital (Unknown); San Paolo Hospital, University of Milan (Unknown); Örebro University, Sweden (Other); San Bassiano Hospital, Vicenza, Italy (Unknown); ALAMIRI Hospital, SABAH ALAHMAD Urology Center, Kuwait (Unknown); Biruni University Medical School, İstanbul, Turkey (Unknown); Jose R. Reyes Memorial Medical Center, Manila, Philippines. (Unknown); Military Medical Academy, Bulgaria (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other); Renmin Hospital of Wuhan University (Other); Wuhan University (Other); The Jiangxi Provincial People's Hospital (Unknown); Affiliated Hospital of Guangdong Medical University (Other); ZhuHai Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Xiangtan Central Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMU Multicentre RCT
Record Dates: First submitted 2021-10-03; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Kidney Calculi
Keywords: Percutaneous nephrolithotomy; Kidney stones; Efficacy; Safety
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in Group 1 undergo suction mini percutaneous nephrolithotomy (Experimental)
  Interventions: Procedure: suction mini percutaneous nephrolithotomy
- Patients in Group 2 undergo standard percutaneous nephrolithotomy (Experimental)
  Interventions: Procedure: standard percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: suction mini percutaneous nephrolithotomy — 18Fr suction sheath (Weili, China) was inserted, and 12Fr mini-nephroscope was used, kidney stones was fragmented by pneumatic lithotriptor (LithoClast Master, Switzerland) or Ho:YAG laser（0.8-1.0W*20-30Hz）, and stone fragments was sucked out with the suction sheath.
  Arms: Patients in Group 1 undergo suction mini percutaneous nephrolithotomy
Procedure: standard percutaneous nephrolithotomy — 24-30Fr sheath was inserted, and 20Fr nephroscope (Richard Wolf, Germany) was used, kidney stones was disintegrated and sucked out by ultrasonic-lithotripter (LithoClast Master, EMS, Switzerland or ShockPluse-SE, Olympus).
  Arms: Patients in Group 2 undergo standard percutaneous nephrolithotomy

SUMMARY:
Percutaneous nephrolithotomy (PCNL) was the first line choice for the management of renal calculi larger than 20 mm. A relative large tract of 24-30Fr was widely used in standard PCNL (sPCNL), which was believed to bring tract-related bleeding. In order to reduce the risk of tract-related bleeding, Chinese urologists used 18Fr mini-tract in the PCNL procedures, which was well known as minimally invasive percutaneous nephrolithotomy (mini-PCNL). In an international multi-centre randomized controlled trail (RCT) , mini-PCNL and sPCNL was compared in the management of 2-4cm kidney stones, the stone free rate (SFR) in mini-PCNL was equal to that of sPCNL. However, since the tract was smaller, the postoperative pain in mini-PCNL was less, the postoperative recovery was faster, and the hospital stay was shorter. Recently, professor Guohua Zeng developed enhanced super-mini-PCNL (eSMP) technique. When compared to traditional mini-PCNL, suction mini-PCNL using 18Fr suction sheath increased the stone removal efficiency and reduced the renal pelvic pressure. While in the present regard, whether suction mini-PCNL play an more efficent and safe role in the management of 2-4cm kidney stones was worthy of further study.

So, the investigators would like to have an international multi-centre RCT to certify our hypothesis.

DETAILED DESCRIPTION:
To certify the efficency and safety of suction mini-PCNL for the management of 2-4cm kidney stones, an international multi-centre RCT was conducted with the comparision of suction mini-PCNL and sPCNL. Investigators plan to do an international multi-centre randomized controlled trial (RCT).

There are 22 hospitals included in this study, including The First Affiliated Hospital of Guangzhou Medical University, Aceves of Wake Forest University Medical Center, University College London Hospital, San Paolo Hospital, University of Milan, Örebro University, San Bassiano Hospital, Vicenza, Italy, ALAMIRI Hospital, SABAH ALAHMAD Urology Center, Kuwait, Biruni University Medical School, İstanbul, Turkey, Jose R. Reyes Memorial Medical Center, Manila, Philippines, Military Medical Academy, The First Affiliated Hospital of Anhui Medical University, The First Affiliated Hospital of Chongqing Medical University, Affiliated Hospital of Zunyi Medical University, The First Affiliated Hospital of Nanchang University, Renmin Hospital of Wuhan University, Xiangtan Central Hospital, Zhongnan Hospital of Wuhan University, The Jiangxi Provincial People's Hospital, Affiliated Hospital of Guangdong Medical University, The First people's Hospital of Foshan, Zhuhai people's Hospital, Nanxishan Hospital of Guangxi Zhuang Autonomous Region.

The primary study endpoints were stone free rate (SFR) and operation time, while the secondary study endpoints were lithotripsy time, hemoglobin drop, transfusion, postoperative fever and other complications, postoperative pain and hospital stay, etc.

This study will be started at August,2021 and ended at August ,2023.

The reported SFR following suction mini-PCNL and sPCNL was 83% and 86%，respectively. The hypothesis was that, the SFR following suction mini-PCNL was higher, or at least not lower than sPCNL. As a bilateral test, α=0.05, test efficiency 1-β=80%, the minimum sample size of each group was determined as n=437. When considered the unfavorable factors, such as withdrawal, n=480 in each group was required, thus the sample size would be 960. In the alternative plan, the sample size was calculated based on the operation time. The reported operation time of suction mini-PCNL and sPCNL for the management of 2-4 cm kidney stones was 45±10 and 35±10 min, respectively. The hypothesis was that, the operation time of suction mini-PCNL was not significantly longer than that of sPCNL. As a bilateral test, α=0.05, the test efficiency 1-β =80%, the non-inferiority test cutoff value for comparing two groups of means was taken as 12, n=310 was calculated for each group.

The sample demand in the second plan was lower than the first plan according to SFR, thus the sample size was finally determined as 960.

The central randomized allocation method was adopted to arrange cases to the sub-centrres. According to the previous daily PCNL procedure volume in each centre, the number of cases in each centre was matched according to the proportion. Ethics committee approval was obtained at each site and informed consent was taken from each patient. A balanced randomization method was used to generate a random number table to each package, so as to ensure a well balance in each centre.

Quality control A standard operating procedure (SOP) was made and approved by the principal investigator of each center. Routine monitoring visits to all centers were carried out every month.

Patients received standard preoperative evaluation, including detailed medical history, physical examination, compete blood count, urinary analysis, midstream urine culture, serum creatinine, electrolyte biochemical tests, coagulation profiles, blood-borne disease screening, non-contrast CT, plain radiography (kidney ureter bladder, KUB), plain chest radiograph, electrocardiogram etc.

Patients with positive preoperative urine culture should be treated with suitable antibiotics based on the culture sensitivity result for at least 7d before standard-PCNL/suction mini-PCNL. Patients who have negative urine culture should receive a single dose of broad spectrum antibiotic prophylaxis in 30mins prior to the procedure.

The potential patients were recruited 3 day before the operation, and the detailed study protocol, the rights and interests of the subjects were informed. Finally, the patients who obtained the written informed consent were enrolled into the present study. The choice of operation mode was based on the corresponding number from the random number table at the time of patients signed the consent, "0" as the standard-PCNL group, "1" as the suction mini- PCNL group.

All procedures was under general anesthesia. After retrograde ureteral catheterization with a 5Fr open-ended catheter, patients were turned to prone position. Under ultrasonography/X-ray guidance, experienced urologists made the puncture into target calyx with an 18-gauge coaxial needle, then 0.035-inch guide-wire was inserted. Fascial dilators were used for the dilation, and the tract was established 18/24Fr by under fluoroscopy guidance.

For suction mini-PCNL, 18Fr suction sheath (Weili, China) was inserted, and 12Fr mini-nephroscope was used, kidney stones was fragmented by pneumatic lithotriptor (LithoClast Master, Switzerland) or Ho:YAG laser（0.8-1.0W*20-30Hz）, and stone fragments was sucked out with the suction sheath.

For standard-PCNL, 24-30Fr sheath was inserted, and 20Fr nephroscope (Richard Wolf, Germany) was used, kidney stones was disintegrated and sucked out by ultrasonic-lithotripter (LithoClast Master, EMS, Switzerland or ShockPluse-SE, Olympus).

At the later stage of the procedure, fluoroscopy was performed to detect the residual stone. Further attempt was made to remove all stone. Double-J stent and/or nephrostomy tube was inserted. Tubeless PCNL was feasible if there was no residual stones, no bleeding, no collecting system perforation nor no ureteral obstruction.

All the stone fragments was collected and the volume of removing stones was evaluated. Stone compositon analysis was obtained. Complete blood count, electrolyte biochemical tests, were performed at 8:00 the next morning after surgery. KUB was required on the 2nd postoperative day to evaluate the stone, stent and tube status. If the stones was completely removed, no additional procedures was needed, no severe bleeding was noted, the nephrostomy tube was removed and patients were discharged. If the residual fragments was≧ 4mm, any information concerning needs for auxiliary treatment should be recorded, including the size of residual stones, the auxiliary treatment and finial outcome. NCCT was requirted to evaluate the final SFR on postoperative one month.

Data collection and definitions of parameters The characteristics of patients and clinical outcomes were recorded according to the pre-established case report form (CRF). Surgical outcomes were predicted preoperatively according to the S·T·O·N·E nephrolithometry. Puncture guidance（Sonography/X ray/combination）, tract location（lower, middle, upper pole and supracostal or subracostal）, tract number, lithotripsy tool, tube and setnt (nephrostomy tube, JJ stent or tubeless). Operation time was defined as the time from puncture to the placement of the nephrostomy tube. Lithotripsy time was defined as the time for lithotripsy only. Hospital stay was defined as days between the surgery date and discharge date. Bruggrmann Comfort Scale (range: 0-5): 0, persistent pain; 1, severe pain while deep breathing or coughing; 2, mild pain while deep breathing or coughing; 3, no pain while deep breathing; 4, no pain while coughing. (Ren C et al. Medicine (Baltimore). 2015 Aug;94(32):e1348.). Visual Analogue Scale (range: 1-10): 0, no pain; 1-3, mild; 4-6, moderate; 7-9, severe; 10, excruciating pain. (Reed MD, Van Nostran W. J Clin Pharmacol. 2014 Mar;54(3):241-4.). Postoperative fever was defined as armpit temperature≥38℃. SIRS was diagnosed in patients who met two or more of the following clinical findings: ① body temperature higher than 38℃ or lower than 36℃;② heart rate higher than 90 beats per minute; ③ respiratory rate greater than 20 breaths per minute or PaCO2 less than 32mm Hg; ④ a white blood cell count higher than 12,000 per mm 3 or lower than 4,000 per mm3. Urosepsis was diagnosed with SOFA scores. Complications of all patients were recorded according to modified Clavien classification system.

Statistical Package for Social Sciences (SPSS) 22.0 was used for statistical analysis. Continuous data was recorded as mean ± standard deviation. Normally distributed data was analyzed with Student's t test, while non-normally distributed data was analyzed with Mann-Whitney U test. Categorical data was reported as n (%), and compared with the χ2 test or Wilcoxon rank sum test. p < 0.05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients consent for percutaneous renal stone removal.
2. Kidney stones 2-4cm.
3. Aged 18-70 years.
4. Normal renal function.
5. ASA scoreⅠ-Ⅱ.

Exclusion Criteria:

1. Severe cardiopulmonary dysfunction or cardiopathy.
2. Coagulation dysfunction.
3. Pyonephrosis or severe acute infection.
4. Transplanted kidney, solitary kidney, horseshoe kidney, urinary diversion, urethra deformity.
5. Other procedure was required in the same session of operation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate (SFR) | 1 month after removing the pigtail stent
  2mm Non-contrast CT is obtained for all patients at one month after removing the pigtail stent to evaluate the final SFR. Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were definded as ≤ 4mm, asymptomatic, non-obstructive and non-infectious stone particles.
Operation time | the time from puncture to the placement of the nephrostomy tube
  Operation time was defined as the time from puncture to the placement of the nephrostomy tube.

SECONDARY OUTCOMES:
Lithotripsy time | the time for lithotripsy only
  Lithotripsy time was defined as the time for lithotripsy only.
Postoperative fever and other complications | intraoperatively or ≤ 1month postoperatively
  Postoperative fever was defined as armpit temperature≥38℃. Complications is defined as any adverse event occurred intraoperatively or ≤ 1month postoperatively, including systemic inflammatory response syndrome (SIRS), urosepsis and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, Ph.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Zeng G, Cai C, Duan X, Xu X, Mao H, Li X, Nie Y, Xie J, Li J, Lu J, Zou X, Mo J, Li C, Li J, Wang W, Yu Y, Fei X, Gu X, Chen J, Kong X, Pang J, Zhu W, Zhao Z, Wu W, Sun H, Liu Y, la Rosette J. Mini Percutaneous Nephrolithotomy Is a Noninferior Modality to Standard Percutaneous Nephrolithotomy for the Management of 20-40mm Renal Calculi: A Multicenter Randomized Controlled Trial. Eur Urol. 2021 Jan;79(1):114-121. doi: 10.1016/j.eururo.2020.09.026. Epub 2020 Sep 29. PMID 32994063
- [Result] Zhong W, Wen J, Peng L, Zeng G. Enhanced super-mini-PCNL (eSMP): low renal pelvic pressure and high stone removal efficiency in a prospective randomized controlled trial. World J Urol. 2021 Mar;39(3):929-934. doi: 10.1007/s00345-020-03263-3. Epub 2020 May 26. PMID 32458093